CLINICAL TRIAL: NCT00566878
Title: A Sub-Registry to Determine the Presence of Alglucosidase Alfa in Breast Milk From Women With Pompe Disease Treated With Alglucosidase Alfa.
Brief Title: Pompe Lactation Sub-Registry
Status: Completed | Type: Observational
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: AGLU03406; LTS13972 (Other: Sanofi)
Record Dates: First submitted 2007-12-01; First posted 2007-12-04 (Estimated); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Glycogen Storage Disease; Pompe Disease
Keywords: Glycogen Storage Disease; GSD-II; Pompe Disease; Pompe Disease (Late-Onset); Acid Maltase Deficiency Disease; Glycogenosis II
MeSH Terms: conditions — Glycogen Storage Disease; Glycogen Storage Disease Type II | interventions — GAA protein, human

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: alglucosidase alfa — At least one infusion of alglucosidase alfa post partum
  Other Names: Myozyme; Lumizyme

SUMMARY:
The objective is to determine if alglucosidase alfa is present in breast milk from mothers with Pompe Disease being treated with alglucosidase alfa and to measure breast milk production and composition in women with Pompe Disease who receive alglucosidase alfa.

ELIGIBILITY:
Inclusion Criteria:

* Must be enrolled in Pompe Registry (NCT00231400)
* Must be pregnant and intend to breast-feed or be currently lactating and receive at least one infusion of alglucosidase alfa while lactating
* Provide a signed Patient Information and Authorization form to participate in the sub-registry prior to any sub-registry-related assessments are performed
* Agree to adhere to the sub-registry guidelines for antibody testing and recommended schedule of assessments.

Exclusion Criteria:

* Patients will be excluded from this sub-registry if they have received an investigational drug (excluding alglucosidase alfa in regions where alglucosidase alfa is not commercially available) within 30 days prior to Visit 1 breast milk collection

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Females diagnosed with Pompe Disease and Lactating
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2012-03-31 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
alglucosidase alfa accumulation in immature (1-3 months post partum) or mature (4-6 months post partum) breast milk sample from mothers with Pompe disease who are being treated with alglucosidase alfa. | 6 Months
breast milk production and composition in women with Pompe disease who receive alglucosidase alfa | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (2):
- United States (2):
  - Registry participation is worldwide. Facilities not yet active may enroll upon identification of a patient, Cambridge, Massachusetts
  - Grand Rapids, Michigan